CLINICAL TRIAL: NCT02258945
Title: Eating Behaviours, Quality of Life and Cardiometabolic Risks in Adults With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion Therapy - A Cross-Sectional Study
Brief Title: CSII in Type 1 Diabetes: Diet, Quality of Life & Cardiometabolic Risks - A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Mr Richard Webb, Postgraduate Research Student, Liverpool John Moores University
Other Study IDs: 13/NW/0122-2
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; CSII; Continuous subcutaneous insulin infusion; Insulin pump; Nutrition; Eating behaviours; Quality of life; Cardiometabolic risks; Liverpool; NHS; Metabolomics; Observational; Lipoproteins; Lipids; Food; Food diary; Cross-Sectional
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Plasma will be retained for use by the research team during the study. After the study remaining samples will be destroyed in accordance with the Human Tissue Authority Code of Practice.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continuous Subcutaneous Insulin Infusion: This group will consist of patients with Type 1 diabetes using continuous subcutaneous insulin infusion therapy.
- Multiple Daily Injections: This group will consist of patients with Type 1 diabetes using multiple daily injection therapy.

SUMMARY:
Glycaemic control is an important aspect of Type 1 diabetes (T1D) management for diabetologists and patients alike. Evidence suggests continuous subcutaneous insulin infusion (CSII) is an effective method of achieving this. Among the advantages of CSII is the opportunity for patients to potentially discard relatively inflexible mealtimes and carbohydrate requirements imposed by other regimes such as multiple daily injections (MDI). There are also reported improvements in quality of life. Furthermore, in patients with good glycaemic control, such as those often assisted by CSII, various qualitative atherogenic lipid abnormalities may exist, despite the presence of a normal quantitative lipid profile; potentially leading to increased cardiometabolic risks. Literature examining the eating behaviours, quality of life and cardiometabolic risks of CSII patients over time after commencement of the therapy is sparse, frequently dated and worthy of further research.

DETAILED DESCRIPTION:
Continuous subcutaneous insulin infusion (CSII) is a therapy for patients with Type-1 diabetes mellitus involving insulin administration via electronic pump. CSII has been shown to reduce HbA1c levels and improve blood sugar control and the continuous, unobtrusive insulin delivery may potentially allow patients increased dietary flexibility and quality of life. However, despite these claims investigatory literature is sparse. This study will clarify whether adult CSII patients experience eating behaviour and quality of life alterations compared to patients using multiple daily injection (MDI) therapy. This is important as differences may be associated with cardiometabolic risk variations; which will also be investigated.

Participants will be a combination of adults with Type-1 diabetes invited from diabetes clinics at the Royal Liverpool University Hospital who are a) have been using CSII for over 1 year or b) have Type 1 diabetes but have never used CSII, have no current plans to use CSII and are presently using MDI therapy.

Following ethical consent participants will be asked to complete one food frequency questionnaire (FFQ) and one quality of life (QOL) questionnaire. A subgroup of these participants (approximately 10 CSII users and 10 MDI users) will then be asked to take part in one interview to investigate quality of life and complete a food diary to explore eating behaviours. All participants consenting to the cross-sectional arm of the study will also be asked to provide an extra volume of blood for analysis. This will be taken at the same time and in addition to their regular diagnostic sample, however where this is unfeasible extra occasional appointments may be needed. (Please be aware that the interview, food diary and blood sample are all optional and that the minimum requirement for participation in the study is the completion of the FFQ and the QOL questionnaires). Results will be compared with existing patient medical records, which will also be analysed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must reside in Liverpool or the surrounding areas.
* Patients must be ages over 18
* Patients must have Type 1 diabetes
* Patients must be using or pending the supply of an insulin pump.
* Patients who have been using either continuous subcutaneous insulin infusion or multiple daily injections for over a year.

Exclusion Criteria:

* Patients must not live outside of Liverpool and the surrounding areas.
* Patients must not be aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Diabetes Centre from the Royal Liverpool and Broadgreen Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Eating behaviours of adult patients with Type 1 diabetes using continuous subcutaneous insulin infusion therapy measured using food diaries and food surveys. | 0 Months
  The primary outcome will be measured at one time point only (due to the cross-sectional nature of the study) using a combination of food frequency questionnaires and food diaries. It is anticipated that all measurements will be taken between April 2014 and December 2014.

SECONDARY OUTCOMES:
Quality of life of adults with Type 1 diabetes who are using insulin pump therapy. | 0 Months
  Quality of life will be assessed at one time point only (due to the nature of the cross-sectional study design) using a combination of semi-structured interviews and quality of life questionnaires.
Cardiometabolic risks of adult patients with Type 1 diabetes who are using insulin pump therapy. | 0 Months
  Cardiometabolic risks will be measured by accessing patient's medical records and taking a sample blood which will be analysed for lipoprotein subfractions, apolipoproteins (A1, A2 and B), HDL, LDL, NEFA, triglycerides and total cholesterol. Metabolomics analysis will also be carried out on collected plasma samples with a focus on both previously identified markers of cardiovascular disease and novel biomarkers. Data will be collected at one time point only (due to the nature of the cross-sectional study design).

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Webb, BA, Principal Investigator — Liverpool John Moores University
Locations (1):
- Royal Liverpool and Broadgreen University Hospital, Liverpool, Merseyside, United Kingdom